CLINICAL TRIAL: NCT04897828
Title: REtrospective Analysis on the Use of COvered Stents for the Treatment of the Dysfunctional Vascular Access
Acronym: RECOVA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital of Patras (Other)
Responsible Party: Principal Investigator, Panagiotis Kitrou, Assistant Porfessor in Interventional Radiology, University Hospital of Patras
Other Study IDs: UHPatras
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Study Focuses on the Use of Covered Stents (Stent Grafts) for the Treatment of Dysfunctional Vascular Access of Hemodialysis Patients
Keywords: covered stent; vascular access; dialysis; arteriovenous fitula; arteriovenous graft

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Covered Stent Group: Patients with a dysfunctional hemodialysis vascular access undergoing treatment procedure using a covered stent (stent graft).
  Interventions: Device: Covered Stent placement

INTERVENTIONS:
Device: Covered Stent placement — Covered stent placement for the treatment of dysfunctional vascular access of hemodialysis patients
  Other Names: Stent placement; Stent Graft placement; Vascular Access intervention

SUMMARY:
This will be a multi-center, multi-national, investigator-initiated and lead, retrospective analysis assessing the safety and the clinical use of covered stents for the treatment of dysfunctional vascular access.

DETAILED DESCRIPTION:
This will be a multi-center, multi-national, investigator initiated and lead retrospective analysis assessing the safety and the clinical use of covered stents for the treatment of the dysfunctional vascular access.

There are no limitations on the type of covered stent use, the reason, or the length of the treatment area. The only limitations are the one owed to covered stent diameter and that patients included in the study should be treated for only one treatment area.

The criteria for inclusion, the outcome measures and the variables that should be recorded are listed below.

There is also no limitation if data has been previously published in another study, however data as part of an ongoing study, or of a study in press cannot be submitted.

Due to previous experience from similar studies it is known that it will be difficult to have data available for all re-interventions. Thus, study will focus on primary patency and safety. Nevertheless, centers should provide data regarding circuit survival (thrombosis, abandonment, surgical revision, patient's death). Terms and definitions of outcome measures are provided below.

Study's final follow-up date is March 31st, 2021. Patient should have a minimum follow-up of 6 months to be included in the study at that timepoint, unless circuit is no longer in use (thrombosis, abandonment, surgical revision, patient's death).

If a scientific committee's approval is needed for the data collection, it is the center's responsibility to acquire it. If this is waived due to the nature of the study, this should also be stated.

A large number of data will be recorded so hopefully, a lot of meaningful evidence will come up from this effort. As seen below, situations out of those allowed in the instructions for use for covered stents are included (ruptures, pseudoaneurysms, cannulation zone placement etc).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <80 years
* Patient on Dialysis with an Arteriovenous Fistula (AVF) or Graft (AVG)
* Clinical Signs of Vascular Access Dysfunction or presence of a Pseudoaneurysm or Intraprocedural Vessel Rupture
* Use of Covered Stent(s) for treatment
* Minimum follow-up: 6 months

Exclusion Criteria:

* >1 treatment areas included per procedure
* Covered Stent not available in the market any more

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that received covered stent treatment for their dysfunctional hemodialysis vascular access at the different centers that will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness: Clinically assessed intervention-free period of the treated segment | 6 months
  A dialysis access circuit with no need for clinically driven treatment area repeat intervention for symptom recurrence and angiographic verification of the presence of stenosis at the treatment area.
Safety: Procedural Complications | 30 days
  Procedure-related Minor Complications No therapy, no consequence Nominal therapy, no consequence; includes overnight admission for observation only
  Procedure-related Major Complications Require therapy, minor hospitalization (<48 hours). Require major therapy, unplanned increase in level of care, Prolonged hospitalization (>48 hours). Permanent adverse sequelae Death

SECONDARY OUTCOMES:
Access Circuit Primary Patency | 12 months
  The interval of patency after an endovascular intervention until any repeat intervention of the access circuit.
Postintervention assisted primary patency | 12 months
  The interval of patency after the endovascular intervention until dialysis circuit thrombosis or a surgical intervention of the access circuit. Endovascular interventions in a previously treated lesion and a new arterial or venous outflow stenosis or occlusion (excluding access thrombosis) are compatible with assisted primary patency. Assisted primary patency ends with percutaneous thrombolysis/thrombectomy or surgical circuit thrombectomy
Anatomic success | 12 months
  Defined as the resumption of normal hemodialysis for a minimum of at least 1 session following percutaneous intervention.
Clinically assessed intervention-free period of the treated segment | 12 months
  A dialysis access circuit with no need for clinically driven treatment area repeat intervention for symptom recurrence and angiographic verification of the presence of stenosis at the treatment area.

OTHER OUTCOMES:
Exploratory analysis | 12 months
  for identification of independent predictors influencing primary outcome measures.

IPD SHARING:
Plan to Share IPD: No
IPD will be collected from investigator sites and statistical analysis will be performed. Results will be presented to the investigators prior to publication.